CLINICAL TRIAL: NCT03721796
Title: Cancer Treatment Decision-making in the HIV Population: an Observational Study of Physician-patient Interactions
Status: Terminated | Type: Observational
Why Stopped: study design changed due to COVID-19
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00101102; CA228631 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Newly Diagnosed Cancer Patients Who Are HIV Positive and Their Treating Oncologist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm 1 Physician/APP: Surgical, medical, and radiation oncologists and/or Advanced Practice Provider (APP)
  Interventions: Other: Audio recording of initial consultation and debriefing interviews.
- Arm 2 Patients: For each participating oncologist, we will may enroll up to three adult cancer patients presenting for consultation, since certain disease sites have a higher incidence in the HIV population.
  Interventions: Other: Audio recording of initial consultation and debriefing interviews.

INTERVENTIONS:
Other: Audio recording of initial consultation and debriefing interviews. — Semi-structured debriefing interviews with participating oncologists and HIV-infected newly diagnosed cancer patients will follow the initial encounter. Interviews will be conducted over 45-60 minutes and will be semi-structured with open-ended questions to allow the interviewee to direct the flow of the conversation.

SUMMARY:
This is a prospective, qualitative study consisting of observation and audio recording of the initial physician-patient consultations in newly diagnosed cancer patients occurring at the Duke University Medical Center (DUMC). Semi-structured debriefing interviews with participating oncologists and patients will follow the initial encounter.

DETAILED DESCRIPTION:
The purpose of this research study is to examine oncologist and patients communication and how patient participation in shared decision-making may impact cancer treatment. Patients who are HIV positive and newly diagnosed with cancer and their treating oncologist may voluntarily participate in this study. The study team will record and observe the initial consultation visit between the patient and treating oncologist. Typically, at this visit, specific treatment options for a new cancer are reviewed in detail. Semi-structured debriefing interviews with participating oncologists and patients will follow the initial encounter.

Patient interviews will occur in person or by telephone within 72 hours of the initial consultation. Oncologists will be interviewed in person within one week following the clinical interaction. Clinical interactions at the initial consultation visit and interviews with oncologists will be audio recorded and transcribed. Interviews will be conducted over 45-60 minutes and will be semi-structured with open-ended questions to allow the interviewee to direct the flow of the conversation. A research assistant trained in qualitative research methods will administer interviews.

There are two to three visits: one visit to complete the informed consent process, the recording of the initial consultation visit, and lastly a debriefing interview visit. The debriefing interview may be conducted in person or over the phone.

The following instruments and question probes will assess three main areas of decision-making:

* Physician Rationale for Decision-Making: In debriefing interviews with physicians, research staff will ask how they arrived at their treatment recommendation and what alternatives they entertained. The extent to which medical comorbidities (including HIV) influenced treatment decision-making and what additional information would have been useful in arriving at the treatment recommendation will be assesssed. We will ask physicians what challenges they encountered in communicating treatment options to the patient, how patient preferences influenced treatment recommendations, and their assessment of how likely the patient is to pursue cancer treatment.
* Strength of Physician Treatment Recommendations: The Physician Recommendation Coding System (PhyReCS) is a validated tool to measure the strength of physician recommendations using direct observation of clinical encounters.64 It is a global, 5-point scale ranging from -2 (strong recommendation against treatment) to +2 (strong recommendation for treatment) that captures how physicians portrayed treatment options during the entirety of the clinical appointment. The PhyReCS addresses major limitations with prior physician decision-making research by having the flexibility to capture multiple nuanced recommendations, for example, patients with early stage breast cancer choosing whether to receive breast-conserving therapy (lumpectomy plus radiation) or mastectomy.
* Patient Preferences: In debriefing interviews with patients, we will elicit beliefs and preferences regarding cancer treatment (e.g. self-efficacy, fear of toxicity, financial hardship, challenges with dual management of co-morbidities and cancer, family support. We will ask patients about their understanding of risks, benefits, and alternatives to treatment and their satisfaction with communication regarding cancer management and outcomes. Patients will be asked if they plan to pursue cancer treatment and if so, which elements of physician communication were most influential.

Patient treatment choice will be determined via chart review 6 months after the initial recorded appointment. We will measure concordance between physician recommendation, strength of the physician recommendation (PhyReCS), and patient treatment choice.

ELIGIBILITY:
Patient Inclusion Criteria:

* Adults 18 years or older
* First diagnosis of primary cancer
* Pre-existing diagnosis of HIV
* Signed and dated informed consent

Physician Inclusion Criteria:

* Must be a practicing medical, radiation or surgical oncologist or APP at Duke Health.
* Signed and dated informed consent

Patient Exclusion Criteria:

* Non-English speaking
* Prior diagnosis of cancer

Physician/APP Exclusion Criteria:

-None applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncologists Newly diagnosed cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Percentage of concordance between physician recommendation and patient treatment decision using the The Physician Recommendation Coding System ( PhyReCS) tool. | 3 years
  The Physician Recommendation Coding System (PhyReCS) is a validated tool to measure the strength of physician recommendations using direct observation of clinical encounters. It is a global, 5-point scale ranging from -2 (strong recommendation against treatment) to +2 (strong recommendation for treatment) that captures how physicians portrayed treatment options during the entirety of the clinical appointment. The PhyReCS addresses major limitations with prior physician decision-making research by having the flexibility to capture multiple nuanced recommendations, for example, patients with early stage breast cancer choosing whether to receive breast-conserving therapy (lumpectomy plus radiation) or mastectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Gita Suneja, MD PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Henry V, Stephens MJ, Galyean P, Young J, Zickmund S, Knettel BA, Bartlett J, Watt MH, Pollak KI, Ubel PA, Fagerlin A, Suneja G. Improving Cancer Care for People Living With HIV: A Qualitative Study of Provider Knowledge, Attitudes, and Practice. Int J Radiat Oncol Biol Phys. 2023 May 1;116(1):60-67. doi: 10.1016/j.ijrobp.2023.01.045. Epub 2023 Jan 29. PMID 36724857